CLINICAL TRIAL: NCT02320773
Title: Non-Interventional Study Assessing Quality of Life, Treatment Satisfaction, Resource Utilisation, and Persistence With Treatment in Overactive Bladder (OAB) Patients Prescribed Betmiga® - A Multicenter Non-interventional Post Authorisation Study (PAS)
Brief Title: A Prospective Non-interventional Study in Overactive Bladder (OAB) Patients Prescribed Betmiga® as Part of Routine Clinical Practice
Acronym: BELIEVE
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 178-MA-1002
Record Dates: First submitted 2014-11-17; First posted 2014-12-19 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Urgency Incontinence; Urinary Bladder Overactive; Overactive Bladder; Urologic Diseases; Urinary Bladder Diseases
Keywords: Overactive Bladder; Quality of Life; Betanis®; Betmiga®; Observational; Myrbetriq®
MeSH Terms: conditions — Urinary Bladder, Overactive; Urologic Diseases; Urinary Bladder Diseases | interventions — mirabegron

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1. OAB patients taking Betmiga®: OAB patients whose physician has made the decision to prescribe Betmiga® as part of routine clinical practice and who are about to start treatment
  Interventions: Drug: Betmiga®

INTERVENTIONS:
Drug: Betmiga® — Oral
  Other Names: YM178; Mirabegron; Myrbetriq®; Betanis®

SUMMARY:
A study to understand the impact of Betmiga® on patients quality of life, satisfaction with treatment, how long patients remain on treatment, patterns of healthcare resource utilisation, and safety as prescribed by the physicians in routine clinical practice.

DETAILED DESCRIPTION:
Single arm, hybrid model study, observing patients on Betmiga under conditions of routine clinical practice, with some element of retrospective data collection 2 years prior to enrolment of the study

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with OAB symptoms at Visit 1 of this study. OAB is defined by the International Urogynecological Association (IUGA)/International Continence Society (ICS) 2010 joint report as urinary urgency, with or without urinary incontinence, usually with frequency and nocturia, with no proven infection or other obvious pathology.
* Patients whose physician has made the decision to prescribe Betmiga® as part of routine clinical practice and who are about to start treatment.

Exclusion Criteria:

* Patients who are currently taking Betmiga®.
* Contraindication(s) as per the Betmiga® Summary of Product Characteristics (SPC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Secondary care centers
Sampling Method: Probability Sample
Enrollment: 863 (Actual)
Dates: Start 2014-11-25 (Actual); Primary Completion 2016-07-27 (Actual); Study Completion 2016-07-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline in QoL based on the OAB-q subscales | Baseline up to 12 months post-baseline
  Quality of life (QoL) based on the Overactive bladder questionnaire (OAB-q) subscales

SECONDARY OUTCOMES:
Change from baseline in patient treatment satisfaction based on TS-VAS | Baseline up to 12 months post-baseline
  Based on Treatment Satisfaction Visual Analogue Scale (TS-VAS)
Change from baseline in QoL based on the EQ-5D-5L subscales and WPAI:SHP | Baseline up to 12 months post-baseline
  QoL based on Work Productivity Activity Index:Specific Health Problem (WPAI:SHP) and EUROQOL 5-DIMENSIONS (EQ5D)
Summary of utilisation of healthcare resources related to the management of OAB | From enrollment to end of study (up to 12 months)
  Overactive bladder (OAB) healthcare resources are captured by the investigator and include: healthcare visits, medical interventions, number of incontinence pads used in last 7 days, invasive/surgical treatments of OAB symptoms and any other investigations of OAB (including clinical interpretation if available)
Frequency summary of disease progression | From enrollment to end of study (up to 12 months
  Disease progression is defined by occurrence of invasive/surgical treatment of OAB symptoms during the study. Overactive Bladder (OAB) treatments include e.g. Botulinum toxin type A, Sacral Neural Stimulation (SNS), Percutaneous tibial nerve stimulation (PTNS)
Change from baseline in incontinence status during the study | Baseline up to 12 months post-baseline
Safety assessed by recording of AEs and ADRs during the study | From enrollment to end of study (up to 12 months)
  Adverse Events (AEs), Adverse Drug Reaction (ADR)
Summary of prescription status to assess treatment patterns and persistence with treatment | Baseline up to 12 months post-baseline
  This composite summary includes the following items:
  * Number and percentage of patients who switched treatment, and to what treatment they were switched.
  * Number and percentage of patients who stopped treatment and reasons associated with discontinuation.
  * Number of treatment days on current treatment.
  * Time from treatment initiation to discontinuation or switching to another treatment.
  * Time from treatment initiation to prescription of additional oral OAB treatment and reasons for combination treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs Europe, Study Director — Astellas Pharma Europe Ltd.
Locations (60):
- Czechia (7):
  - Site CZ42009 UROMEDA s. r. o., Brno
  - Site CZ42003 Fakultni nemocnice Brno-Bohunice, Brno
  - Site CZ42006 Hospital Kyjov, Kyjov
  - Site CZ42002 Fakultni nemocnice Kralovske Vinohrady, Prague
  - Site CZ42007 MEDICON a.s., Prague
  - Site CZ42008 Oblastni nemocnice Pribram, Příbram
  - Site CZ42004 Krajská nemocnice Tomáše Bati, Zlín
- Denmark (2):
  - Site DK45003 Sygehus Vendsyssel, Frederikshavn, Frederikshavn
  - Site DK45004 Regionshospitalet Herning, Herning
- Greece (11):
  - Site GR30002 University Hospital of Crete, Heraklion, Crete
  - Site GR30009 PGH Laiko, Athens
  - Site GR30001 General Hospital of Athens "Alexandra", Athens
  - Site GR30007 Sismanoglio General Hospital, Athens
  - Site GR30011 General Hospital of Heraklion 'Venizelio-Pananio', Heraklion
  - Site GR30008 University Hospital of Ioannina, Ioannina
  - Site GR30013 University Hospital of Ioannina, Ioannina
  - Site GR30005 University Hospital of Larissa, Larissa
  - Site GR30003 University Hospital of Patras, Pátrai
  - Site GR30006 Papageorgiou General Hospital, Thessaloniki
  - Site GR30012 Papageorgiou General Hospital of Thessaloniki, Thessaloniki
- Ireland (3):
  - Site IE35304 Midland Regional Hospital, Mullingar, Co. Westmeath
  - Site IE35302 Coombe Hospital, Dublin
  - Site IE35303 Kerry General Hospital, Kerry
- Slovakia (7):
  - Site SK42101 Univerzitná nemocnica Bratislava - Kramáre, Bratislava
  - Site SK42106 UROCENTRUM LEVICE, s.r.o., Levice
  - Site SK42102 UROAMB, s.r.o., Liptovský Mikuláš
  - Site SK42104 Urologicka ambulancia, Miramed, sro, Rimavská Sobota
  - Site SK42107 Private Urological Care Center, Trenčín
  - Site SK42103 CMFF, sro, Vranov nad Topľou
  - Site SK42105 ProCare Ziar nad Hronom, Žiar nad Hronom
- Spain (11):
  - Site ES34005 Corporació Sanitaria Parc Taulí, Sabadell, Barcelona
  - Site ES34012 H. de Mendaro, Mendaro, Guipuzcoa
  - Site ES34015 Centro Médico Teknon, Barcelona
  - Site ES34007 Hospital Universitario Vall D'Hebron, Barcelona
  - Site ES34017 Hospital de Mollet, Barcelona
  - Site ES34020 Hospital Universitario Basurto, Bilbao
  - Site ES34009 Hospital Comarcal Santiago Apostol, Burgos
  - Site ES34021 H. de Donostia, Donostia / San Sebastian
  - Site ES34019 Hospital Universitario Lucus Augusti, Lugo
  - Site ES34011 Hospital del Rio Hortega, Valladolid
  - Site ES34010 Policlínico de Vigo, S.A.-POVISA, Vigo
- Site SE46002 Urologkliniken Carlanderska, Gothenburg, Sweden
- United Kingdom (18):
  - Site GB44005 Bradford Royal Infirmary, Bradford
  - Site GB44011 Royal Blackburn Hospital, Burnley
  - Site GB44016 Addenbrookes Hospital, Cambridge
  - Site GB44009 St. Richards Hospital, Chichester
  - Site GB44007 Northampton General Hospital, Cliftonville
  - Site GB44015 University Hospital Coventry, Coventry
  - Site GB44008 Croydon University Hospital, Croydon
  - Site GB44003 Derriford Hospital, Derriford
  - Site GB44019 Northern Devon Healthcare, Devon
  - Site GB44001 Medway Hospital, Gillingham
  - Site GB44004 Southern General Hospital, Glasgow
  - Site GB44013 Hinchingbrooke Hospital, Huntingdon
  - Site GB44010 The Freeman Hospital, Newcastle upon Tyne
  - Site GB44014 The Queen Elizabeth Hospital King's Lynn NHS Trust, Norfolk
  - Site GB44002 The Royal Berkshire Hospital, Reading
  - Site GB44018 Salisbury District Hospital, Salisbury
  - Site GB44017 Sunderland Royal University Hospital, Sunderland
  - Site GB44006 New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Freeman R, Foley S, Rosa Arias J, Vicente E, Grill R, Kachlirova Z, Stari A, Huang M, Choudhury N. Mirabegron improves quality-of-life, treatment satisfaction, and persistence in patients with overactive bladder: a multi-center, non-interventional, real-world, 12-month study. Curr Med Res Opin. 2018 May;34(5):785-793. doi: 10.1080/03007995.2017.1419170. Epub 2018 Jan 10. PMID 29254376
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/study.aspx?ID=223